CLINICAL TRIAL: NCT03600688
Title: Transcatheter Repair of Mitral Regurgitation With Cardioband System Post Market Study:A European Prospective, Multicenter Study to Assess Transcatheter Mitral Valve Repair With Edwards Cardioband System in Patients With Symptomatic MR
Brief Title: Edwards Cardioband European Post-Market Study, MiBAND
Acronym: MiBAND
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-10
Record Dates: First submitted 2018-06-15; First posted 2018-07-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Mitral Regurgitation; Mitral Insufficiency; Mitral Repair; Mitral Valve; Annuloplasty; Edwards Cardioband
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Edwards Cardioband System — Transcatheter mitral valve repair

SUMMARY:
To demonstrate reduction of MR with durable performance and im-provements in functional status

DETAILED DESCRIPTION:
MiBAND is a prospective, single arm, European post-market study to assess the safety and efficacy of the Edwards Cardioband system. Patients will be followed up at 30D, 6months, 1, 2 and 3 years.

ELIGIBILITY:
Main Inclusion Criteria:

* Age ≥ 18 years;
* MR (≥ 2+ by echocardiography);
* Patient is eligible to receive the Edwards Cardioband Mitral System

Main Exclusion Criteria:

* Active bacterial endocarditis
* Severe organic lesions with retracted chordae or congenital mal-formations with lack of valvular tissue
* Heavily calcified annulus or leaflets
* Patients in whom transesophageal echocardiography is contraindicated
* Patients who cannot tolerate an anticoagulation/antiplatelet regimen
* Patients with known severe reaction to contrast agents that cannot be adequately pre-medicated.
* Pre-existing prosthetic heart valve or annuloplasty in the Mitral position
* Life expectancy of less than twelve months
* Patient is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic patients with mitral regurgitation (MR).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-06-06 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedure Success at discharge | Hospital discharge; approximately 2-8 days post-procedure
  Reduction in Severity of Mitral Regurgitation at discharge

SECONDARY OUTCOMES:
Procedure Success | 30 days, 6months, 1, 2 and 3 years
  Reduction in Severity of Mitral Regurgitation
Major Adverse Events Rate | 30 days, 6months, 1, 2 and 3 years
  Rate of Major Adverse Events
Change in Quality Of Life-KCCQ | 30 days, 6 months, 1, 2 and 3 years
  Improvements in Quality Of Life as assessed by KCCQ
Change in Quality Of Life-EQ-5D-5L | 30 days, 6 months, 1, 2 and 3 years
  Improvements in Quality Of Life as assessed by EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Baldus, MD, Principal Investigator — Herzzentrum UniKlinik Köln
Locations (17):
- Germany (11):
  - Herz- und Diabeteszentrum NRW Bad Oeynhausen, Bad Oeynhausen
  - Berlin Charité - Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Herzzentrum UniKlinik Köln, Cologne
  - Herzzentrum Universitästklinik Dresden, Dresden
  - Düsseldorf University Hospital, Düsseldorf
  - Goethe-University Frankfurt - Surgery Center, Frankfurt am Main
  - Universitätsmedizin Göttingen, Göttingen
  - Asklepios Klinik St Georg, Hamburg
  - Universtitätsmedizin Mainz, Mainz
  - Universitätsklinikum Münster, Münster
- Italy (5):
  - Policlinico Vittorio-Emanuelle, Catania
  - Ospedale del Cuore G. Pasquinucci - Fondazione Toscana Gabreile Monasterio, Massa
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Policlinico San Donato, San Donato Milanese
- University Hospital Zürich, Zurich, Switzerland